CLINICAL TRIAL: NCT04326933
Title: Effects of Tyrosine Kinase Inhibitors on Liver Enzymes and Electrolytes in Relation to Hematologic Response in Patients With Chronic Phase Chronic Meyloid Leukemia: Assiut University Hospital Insight
Brief Title: Effects of Tyrosine Kinase Inhibitors on Liver Enzymes and Electrolytes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Mahmoud, Principal investigator, Assiut University
Other Study IDs: TKI In CML
Record Dates: First submitted 2019-11-21; First posted 2020-03-30 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Patients Diagnosed as Chronic Meyloid Leukemia
MeSH Terms: interventions — Tyrosine Kinase Inhibitors; Imatinib Mesylate; nilotinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tyrosine kinase Inhibitors (Imatinib & Nilotinib) — Administration of tyrosine kinase inhibitors (Imatinib in a dose of 400mg/day & Nilotinib in adose of 600mg/day)
  Other Names: Glivic & Tasigna

SUMMARY:
Determine the effects of tyrosine kinase Inhibitors on liver enzymes and electrolytes in relation to hematologic response in patients with chronic phase chronic meyloid leukemia.. Assiut University Hospital insight..

DETAILED DESCRIPTION:
CML is a myeloproliferative neoplasm with unique biological and clinical features.

CML accounts for 15_20% of newly diagnosed cases of leukemias among adults. CML can present in three clinical phases : chronic phase, accelerated phase and blast phase.

CML is characterized by prodction of a breakpoint cluster region abelson(BCR-ABL) fusion protein with ABL kinase activity. This is due to reciprocal translocation between chromosome 9 and 22.

Imatinib & Nilotinib, an ABL kinase inhibitors, which has revolutionized the CML therapy, are a selective tyrosine kinase inhibitors.

The aim of the study is to determine the changes of liver enzymes and electrolytes in relation to hematologic response during treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with CML
* Chronic phase CML
* Normal hepatic and renal functions

Exclusion Criteria:

* Blastic phase CML
* Accelerated phase CML
* Hepatic & renal impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with chronic phase chronic meyloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Follow up liver enzymes as AST, ALT, ALP and GGT before starting treatment and during the period of treatment by Tyrosine Kinase Inhibitors (Imatinib & Nilotinib). | 6 months
  Changes happen in liver enzymes after a period of treatment by Tyrosine Kinase Inhibitors (Imatinib & Nilotinib) which are assessed by measuring liver enzymes as AST, ALT, ALP, GGT before starting treatment and during the period of treatment and the relation between these changes and the hematologic response to the treatment that is assessed by CBC and BCR-ABL Gene.
Follow up electrolytes as Na, K, Ca and P before starting treatment and during the period of treatment by Tyrosine Kinase Inhibitors (Imatinib & Nilotinib) | 6 months
  Changes happen in electrolytes after a period of treatment by Tyrosine Kinase Inhibitors (Imatinib & Nilotinib) which are assessed by measuring electrolytes levels before starting treatment and during the period of treatment and the relation between these changes and the hematologic response to the treatment that is assessed by CBC and BCR-ABL Gene

CONTACTS AND LOCATIONS:
Overall Officials: Howaida A Nafady, Prof., Principal Investigator — Not affiliated
Locations (1):
- Assiut University Hospital, Asyut, Egypt